CLINICAL TRIAL: NCT04481490
Title: Objective Measure of Physical Activity and Sedentary Behavior During Cardiac Rehabilitation: Are Patients Achieving Recommendations/Guidelines
Brief Title: A Study to Objectively Measure Physical Activity and Sedentary Behavior During Cardiac Rehabilitation
Status: Withdrawn | Type: Observational
Why Stopped: Stopped due to lack of personnel and funding support
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amanda R. Bonikowske, Principal Investigator, Mayo Clinic
Other Study IDs: 20-005866
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Disease; Myocardial Infarction; Cardiac Valve Disease; Coronary Artery Disease
Keywords: cardiac rehabilitation; physical activity; accelerometry; home-based
MeSH Terms: conditions — Heart Diseases; Myocardial Infarction; Heart Valve Diseases; Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Home-based: Cardiac rehabilitation (including exercise training) delivered in a home-based setting, facilitated remotely by Mayo Clinic staff.
- Center-based: Cardiac rehabilitation (including exercise training) delivered in a center-based setting, facilitated in person by Mayo Clinic staff.

SUMMARY:
The purpose of this study is to assess exercise patterns during home-based or center-based cardiac rehabilitation participation.

DETAILED DESCRIPTION:
Participants enrolled in either home-based or center-based cardiac rehabilitation will be instructed to wear an accelerometer device for 7-days at baseline, 4-weeks, 8-weeks, and 12-weeks, to objectively measure their physical activity level during the cardiac rehabilitation program. A questionnaire will also be completed by the participant at baseline and 12-weeks to subjectively measure their physical activity level, based on self-report activities over the previous 7-days.

Enrollment in home-based versus center-based cardiac rehabilitation will be based on the availability of cardiac rehabilitation facilities and/or patient preference. There is no random allocation or assignment to groups by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older.
* Able to provide consent.
* Has a qualifying indication for cardiac rehabilitation and able to participate in cardiac rehabilitation.

Exclusion Criteria:

* Unwilling or unable to participate in cardiac rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with qualifying indication for cardiac rehabilitation (e.g. acute coronary syndrome, myocardial infarction, percutaneous coronary intervention, coronary artery bypass grafting, stable angina, heart failure).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in minutes spent in moderate-vigorous physical activity, measured by accelerometry | Baseline, 4-weeks, 8-weeks, and 12-weeks
  Change in minutes at a moderate-vigorous activity intensity are objectively measured by an accelerometer device that senses movement. The device captures the number of minutes a participant spends in moderate-vigorous activities per day, and will be worn by the participant for 7-days. A higher number of minutes per day indicates a greater physical activity level.

SECONDARY OUTCOMES:
Change in minutes spent in moderate-vigorous physical activity, measured by questionnaire | Baseline, 12-weeks
  Change in minutes at a moderate-vigorous activity intensity are subjectively measured (self-reported) using the International Physical Activity Questionnaire (IPAQ). The IPAQ captures the number of minutes a participant spends in moderate-vigorous activities per day, based on participant's reporting of the previous 7-days. A higher number of minutes per day indicates a greater physical activity level.
Change in minutes spent in inactive (sedentary) behavior, measured by accelerometry. | Baseline, 4-weeks, 8-weeks, and 12-weeks
  Change in minutes spent in inactive (sedentary) behavior, measured by an accelerometer device that senses movement. The device captures the number of minutes a participant spends inactive per day, and will be worn by the participant for 7-days. A higher number of minutes per day of inactive time indicates increased sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Bonikowske, PhD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials